CLINICAL TRIAL: NCT00660023
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety, and Tolerability of Once-Monthly Administration of Intravenous C.E.R.A. for the Maintenance of Haemoglobin Levels in Dialysis Patients With Chronic Renal Anaemia
Brief Title: A Study of Intravenous Mircera in Participants With Chronic Renal Anemia Who Are on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20752; 2006-005621-28
Record Dates: First submitted 2008-04-16; First posted 2008-04-17 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera in Renal Anemia (Experimental): Participants with chronic renal anemia previously treated with ESA therapy will receive intravenous Mircera, also known as continuous erythropoietin receptor activator (CERA), every 4 weeks for a total of 52 weeks in this single-arm study. The first dose will be determined by the dose of ESA received prior to administration of study treatment, and subsequent doses will be adjusted to achieve target Hb concentrations.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Participants will receive intravenous CERA/Mircera every month, with starting dose based on previous ESA therapy. Treatment will continue for 52 weeks.
  Other Names: CERA/Mircera

SUMMARY:
This single-arm study will assess the efficacy and safety of monthly administration of intravenous methoxy polyethylene glycol-epoetin beta (CERA/Mircera) for the maintenance of hemoglobin (Hb) levels in participants on dialysis with chronic renal anemia in routine clinical practice in Hungary. Participants currently receiving maintenance treatment with intravenous epoetin or darbepoetin will receive monthly injections of Mircera, with the starting dose derived from the erythropoiesis-stimulating agent (ESA) dose they had been receiving.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Chronic renal anemia
* Continuous stable intravenous or subcutaneous maintenance epoetin or darbepoetin therapy during previous month
* Regular long-term hemodialysis therapy with the same mode of dialysis for the previous 3 months

Exclusion Criteria:

* Transfusion of red blood cells during previous 2 months
* Poorly controlled hypertension
* Significant acute or chronic bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Hungary (10):
  - Baja
  - Budapest
  - Debrecen
  - Esztergom
  - Keszthely
  - Miskolc
  - Salgótarján
  - Szolnok
  - Vác
  - Zalaegerszeg

REFERENCES:
- [Derived] Locatelli F, Choukroun G, Truman M, Wiggenhauser A, Fliser D. Once-Monthly Continuous Erythropoietin Receptor Activator (C.E.R.A.) in Patients with Hemodialysis-Dependent Chronic Kidney Disease: Pooled Data from Phase III Trials. Adv Ther. 2016 Apr;33(4):610-25. doi: 10.1007/s12325-016-0309-6. Epub 2016 Mar 10. PMID 26965694

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with erythropoiesis-stimulating agent (ESA) therapy received intravenous methoxy polyethylene glycol-epoetin beta (Mircera), also known as continuous erythropoietin receptor activator (CERA), every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 micrograms (mcg) was based upon the dose of ESA received in the week preceding the switch to Mircera/CERA, while subsequent doses were adjusted to maintain hemoglobin (Hb) concentrations within target of 10.0 and 12.0 grams per deciliter (g/dL).
Period: Overall Study
Arm/Group | Mircera in Renal Anemia
Started | 124
Treated | 114
Completed | 95
Not Completed | 29
Not completed — Adverse Event | 2
Not completed — Death | 8
Not completed — Blood Transfusion | 5
Not completed — Renal Transplantation | 3
Not completed — Withdrawal by Subject | 1
Not completed — Missed Pregnancy Test | 1
Not completed — Other Screening Failure | 9

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of Mircera/CERA and for whom data from at least one follow-up assessment were available.
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with ESA therapy received intravenous Mircera/CERA, every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg was based upon the dose of ESA received in the week preceding the switch to Mircera/CERA, while subsequent doses were adjusted to maintain Hb concentrations within target of 10.0 and 12.0 g/dL.
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
Age, Continuous [Median (Full Range); unit: years] | 63.5 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Average Hb Within Plus/Minus (±) 1 g/dL of Reference Hb and Within Target Range During the Efficacy Evaluation Period (EEP)
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to -1). During the EEP (Weeks 18 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with CERA/Mircera. The average Hb during the EEP was calculated per participant and assessed against the reference value. The percentage of participants who had average Hb during the EEP in the target range of 10.0 to 12.0 g/dL and within ±1 g/dL of their individual reference Hb was determined as the primary endpoint. The 95 percent (%) confidence interval (CI) was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Weeks -4, -3, -2, and -1; pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: Per Protocol (PP) Population: All participants from the ITT Population who fulfill inclusion/exclusion criteria per study protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 88
percentage of participants | 72.7 [62.2 to 81.7]

2. Secondary Outcome: Mean Change in Time-Adjusted Hb From Baseline to EEP
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment stability assessment (Weeks -4 to -1). During the EEP (Weeks 18 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with CERA/Mircera. The average Hb during the EEP was calculated per participant and assessed against the reference value. The mean change in Hb value between reference (i.e., "Baseline") Hb and the EEP average Hb was calculated and expressed in g/dL.
Time Frame: At Weeks -4, -3, -2, and -1; pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
g/dL | -0.06 (1.04)

3. Secondary Outcome: Percentage of Participants Whose Hb Remained Within Target Range Throughout the EEP
Description: During the EEP (Weeks 18 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with CERA/Mircera. The percentage of participants who maintained each single Hb measurement in the target range of 10.0 to 12.0 g/dL was determined. The 95% CI was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
percentage of participants | 79.0 [70.3 to 86.0]

4. Secondary Outcome: Mean Time Spent in the Target Range for Hb During the EEP
Description: During the EEP (Weeks 18 to 24), participants provided a total of four blood samples for Hb monitoring while on treatment with CERA/Mircera. Time spent in the target range of 10.0 to 12.0 g/dL was defined as time from first on-target Hb to time of last known on-target Hb, as collected during the EEP. Time spent in the target range was averaged among all participants and expressed in days.
Time Frame: Pre-dose (0 hours) during Weeks 18, 20, 22, and 24
Population: ITT Population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
days | 43.5 (15.64)

5. Secondary Outcome: Mean Dose of Mircera/CERA During the Dose Titration Period (DTP) and EEP
Description: Study drug administration occurred monthly during the DTP (Weeks 0 to 16), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during Week -1. Subsequent doses could be adjusted throughout the study including during the EEP (Weeks 18 to 24) on the basis of Hb levels or other modification criteria. The dose received at each administration visit was averaged among all participants during the DTP and EEP and expressed in mcg.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: ITT Population; the number (n) of participants who received at least one dose during the specific period was used for analysis.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
mcg
  DTP (n=114) | 113 (39.4)
  EEP (n=110) | 100.3 (69.43)

6. Secondary Outcome: Percentage of Participants Who Required Any Dose Adjustment of Mircera/CERA During the DTP and EEP
Description: Study drug administration occurred monthly during the DTP (Weeks 0 to 16), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during Week -1. Subsequent doses could be adjusted throughout the study including during the EEP (Weeks 18 to 24) on the basis of Hb levels or other modification criteria. The percentage of participants who required a dose adjustment for any reason was calculated during the DTP and EEP.
Time Frame: Weeks 0, 4, 8, 12, 16, 20, and 24
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
percentage of participants
  DTP (n=114) | 79.8
  EEP (n=110) | 48.2

7. Secondary Outcome: Number of Participants Receiving Blood Transfusion During the DTP and EEP
Description: The number of participants who received blood transfusion during the DTP (Weeks 0 and 16) and EEP (Weeks 18 to 24) was reported.
Time Frame: Continuously and at every visit from Week 0 (every week until Week 2, thereafter every 2 weeks) through Week 24
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
participants
  DTP (n=114) | 3
  EEP (n=110) | 0

8. Secondary Outcome: Number of Blood Transfusions During the DTP and EEP
Description: The number of blood transfusion during the DTP (Weeks 0 and 16) and EEP (Weeks 18 to 24) was reported.
Time Frame: Continuously and at every visit from Week 0 (every week until Week 2, thereafter every 2 weeks) through Week 24
Population: as for outcome 5
Measure: Number; unit: blood transfusions
Arm/Group | Mircera in Renal Anemia
Number analyzed (Participants) | 114
blood transfusions
  DTP (n=114) | 4
  EEP (n=110) | 0

ADVERSE EVENTS:
Time Frame: Continuously and at every visit from Week -3 (every week until Week 2, every 2 weeks until Week 48) through the final visit at Week 52
Description: Safety Population: All participants who received at least one dose of trial medication and at least one safety follow-up assessment, whether prematurely withdrawn or not.
Groups:
- Mircera in Renal Anemia: Participants with chronic renal anemia who were previously treated with ESA therapy received intravenous Mircera/CERA, every 4 weeks for a total of 52 weeks in this single-arm study. The first dose of 120, 200, or 360 mcg was based upon the dose of ESA in the week preceding the switch to Mircera/CERA, while subsequent doses were adjusted to maintain Hb concentrations within target of 10.0 and 12.0 g/dL.
Arm/Group | Mircera in Renal Anemia
Serious Adverse Events (participants affected / at risk) | 45/114
Other Adverse Events (participants affected / at risk) | 40/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=114)
Haemolysis (Blood and lymphatic system disorders) | 1
Cardiac asthma (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 4
Cardiovascular disorder (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Medical device complication (General disorders) | 2
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Renal cyst infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 1
Haemoglobin decreased (Investigations) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 2
Cerebrovascular disorder (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Cataract operation (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Intermittent claudication (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in Renal Anemia (N=114)
Bronchitis (Infections and infestations) | 8
Muscle spasm (Musculoskeletal and connective tissue disorders) | 9
Hypertension (Vascular disorders) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.